CLINICAL TRIAL: NCT00991601
Title: Ultra Sound Guided Fine Needle Aspiration Cytology (FNAC) of Liver and Pancreas Tumours
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: New ultra sound technology have made this present study design less relevant and force us to change the design of the study.
Sponsor: Herlev Hospital (Other)
Responsible Party: Jakob Burcharth, MD., Herlev Hospital, Department of surgical Gastroenterology
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-KA-05092
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Tumors in Liver; Tumors in Pancreas
Keywords: liver; pancreas; cancer; tumor; FNAC
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- biopsy arm (Experimental): patients with tumors in liver and/or pancreas
  Interventions: Procedure: FNAC (fine needle aspiration cytology)

INTERVENTIONS:
Procedure: FNAC (fine needle aspiration cytology) — UL guided biopsy

SUMMARY:
Patients with tumors in liver or pancreas are randomized to ultrasound (UL)-guided FNAC biopsies with guidance method or UL-guided FNAC biopsies with free-hand method.

ELIGIBILITY:
Inclusion Criteria:

* adult over 18 years
* tumors in liver and/or pancreas

Exclusion Criteria:

* low coagulation factors
* mentally ill patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
quality of obtained biopsy | one year

SECONDARY OUTCOMES:
patients pain and discomfort at procedure | immediately

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Burcharth, MD, Principal Investigator — Herlev Hospital; Bjørn Skjoldbye, MD, Study Director — Herlev Hospital
Locations (1):
- Herlev Hospital, Dk-2730, Herlev, Herlev, Denmark